CLINICAL TRIAL: NCT02333981
Title: Efficacy of Passive Oral Motor Therapy on Drooling in Children With Multiple Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, DIVYA MIDHA, ASSISTANT PROFESSOR, Maharishi Markendeswar University (Deemed to be University)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1234
Record Dates: First submitted 2015-01-01; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Disabilities

ARMS (1):
- Passive oral motor therapy group (Experimental): All the subjects received passive treatment which included light touch, stroking, vibration, tapping, pressure and stretch. All the techniques have been proved to be effective in treating drooling. Relative sterility and hygiene was maintained throughout the procedure as sterilized gloves and napkins were used. The measurement protocol was designed to check effectiveness on drooling in children. The protocol was given for 4 weeks with treatment sessions given 3 times per week and the treatment duration was 30min.12 sessions of oral motor stimulation therapy given during the 4 weeks..
  Interventions: Device: passive oral motor therapy for drooling

INTERVENTIONS:
Device: passive oral motor therapy for drooling — 7 subjects aged 7-19 yrs were taken . All subjects received passive treatment which included light touch, stroking, vibration with (mechanical vibrator), tapping, pressure and stretch. All the techniques have been proved to be effective in treating drooling. Relative sterility and hygiene was maintained throughout the procedure as sterilized gloves and napkins were used. The measurement protocol was designed to check effectiveness on drooling in children. The protocol was given for 4 weeks with treatment sessions given 3 times per week and the treatment duration was 30min.12 sessions of oral motor stimulation therapy given during the 4 weeks..

SUMMARY:
This study was formulated to determine the efficacy of passive oral motor regimen for drooling in children with multiple disabilities. Seven subjects aged 7-19yrs were taken in the study. All the subjects received passive treatment which included light touch, stroking, vibration, tapping, pressure and stretch. All the techniques have been proved to be effective in treating drooling. Relative sterility and hygiene was maintained throughout the procedure as sterilized gloves and napkins were used. The measurement protocol was designed to check effectiveness on drooling in children. The protocol was given for 4 weeks with treatment sessions given 3 times per week and the treatment duration was 30min. Twelve sessions of oral motor stimulation therapy given during the 4 weeks. Thirteen after 4 weeks of treatment, improvement was found in terms of the severity as well. Primary outcome measure taken was Drooling Frequency and Severity rating scale and secondary outcome measure being taken was drool quotient. Pre and post intervention scores of Drooling Frequency and Severity rating scale and drool quotient were taken and data was analyzed using wilcoxon signed rank test .

DETAILED DESCRIPTION:
Title To formulate and see efficacy of passive oral motor regimen for drooling in children with multiple disabilities Background Drooling ranges from mild embarrassment and discomfort for the intellectually intact patient with minimal drooling to gross emotional and physical impairment for the severely affected individual. Drooling produces an unhygienic condition that may be associated with a disagreeable odour. Drooling affects the social and physical wellbeing of children and may represent problems for caregivers. Many persons with severe and profound disabilities exhibit chronic and excessive drooling, which can have unfavourable effects on their socialization and health. Studies have suggested that various treatments like medication, surgery, behaviour modification, myofunctional therapy and oral motor therapy are effective in treating drooling but there is no single protocol developed to treat drooling in children with multiple disabilities. Passive treatment protocol is needed specifically designed for children who are not able to follow commands and on whom various treatment techniques like behaviour modification, over-correction can't be applied. Present study aims to formulate and see the efficacy of passive oral motor regimen for drooling in children with multiple disabilities.

Methodology Seven subjects of age group between 07-19 years were selected out of accessible population.

Informed consent taken from the parents/caregivers.Severity and frequency of drooling accessed (For each subject prior to the study) and Drool Quotient was calculated (For each subject prior to the study). Patient was in sitting position with back fully supported and head in neutral position in their own home. Therapist in standing position in front of the patient.Therapist wore sterilised gloves to ensure that no infection occurs along with change of gloves for every subject. Light touch applied to mid line of lips (3 times, for 5 sec). Maintained pressure applied around lips (3 times for 3 sec). Gentle tapping to the cheeks applied with index finger (8 times each cheek). Quick, gentle stretch applied outward with index and middle finger on middle of upper lip and lower lip (8 times on each lip). Gentle stroke to the cheek applied with index finger from base of nose towards ear. Then returned back to corner of lips (8 times each cheek), repeat on the other side. Gentle stroking applied to area around the lips in a circular manner, from the corner towards the center and to the other corner, then reverse. (4 times each lip). Vibration slowly applied for 10-15 sec each of a) orbicularis oris b) Both sides of larynx from chin to sternal notch c) Under the chin from ear to ear.Quick stretch applied to the masseter muscles (3 times on each side). Stretch pressure applied to vibrated areas, on a) orbicularis oris b) Laryngopharyngeal muscles, both sides. Intra-orally applied light touch to roof of mouth, anteriorly for 3 times. The protocol was given for 4 weeks with treatment sessions given 3 times per week.

.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-19 yrs (male and female)
* Confirmed diagnosis of multiple disability Score of ≤ 3 on drooling severity and frequency scale (indicating moderate to profuse drooling)
* Medication, taken to treat drooling, stopped at least 3 months before start of the study

Exclusion Criteria:

* No History of Previous surgical procedure for saliva control
* Use of drugs that interfere with saliva secretion (anticholinergic and neuroleptic drugs, benzodiazepines)
* Use of oral prosthetic devices
* Tactile hypersensitivity and oral problems like caries, toothache
* Congenital defects like cleft palate
* systemic diseases (bronchial asthma, congenital heart failure, and myasthenia gravis)
* Previous surgical procedures in the oral/nasal cavity interfering with saliva production
* Respiratory dysfunction

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Drooling Frequency and Severity rating scale | 4 weeks

SECONDARY OUTCOMES:
Drool Quotient method | 4 weeks
  METHOD OF ASSESSMENT OF SEVERITY OF DROOLING

CONTACTS AND LOCATIONS:
Overall Officials: DIVYA MIDHA, MPT(NEURO), Principal Investigator — MAHARISHI MARKANDESHWAR UNIVERSITY